CLINICAL TRIAL: NCT01727947
Title: Influence of Sperm With Large Nuclear Vacuoles on the Cycles' Outcomes of Couples Couples Undergoing ICSI
Brief Title: Influence of Sperm With Large Nuclear Vacuole on ICSI Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sapientiae Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: MSOME_SLV
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSOME (Experimental): Couples in which the sperm cells were analysed through MSOME
  Interventions: Other: MSOME

INTERVENTIONS:
Other: MSOME — A total of 200 spermatozoa of each sample will be analyzed under high magnification (x6600) and the incidence of SLV (sperm cells presenting at least one vacuole that occupied > 13% of nuclear area) in each sample will be assessed.

SUMMARY:
Current research on sperm morphology has been directed towards the dysmorphisms of the sperm head. A new technique based on the motile sperm organelle morphology examination (MSOME) allows the detection of sperm with large nuclear vacuoles (SLV). Large nuclear vacuoles are specific sperm alterations observed under high magnification, and their presence has been related to increased DNA fragmentation and denaturation.

DETAILED DESCRIPTION:
A new method for the detailed morphological evaluation of motile spermatozoa in real time, under high magnification, named "motile sperm organellar morphology examination" (MSOME) was developed. This magnification provides an accurate description of spermatozoa abnormalities, particularly the presence of head vacuoles, which is indicative of abnormal chromatin packaging in spermatozoa. However, the influence of sperm with large nuclear vacuoles (SLV) on ART outcomes is still a matter of debate. The goals for this study were to identify whether there is a connection between SLV under high magnification and ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing intracytoplasmic sperm injection (ICSI) as result of male factor or tubal factor or unexplained infertility
* Women with regular menstrual cycles of 25-35 days
* Women with normal basal follicle stimulating hormone (FSH) and luteinizing hormone (LH) levels
* Women with body mass index (BMI) less than 30 kg/m2
* Women with both ovaries and intact uterus

Exclusion Criteria:

* Women with polycystic ovaries syndrome
* Women with endometriosis
* Women with gynaecological/medical disorders
* Couples with any sexually transmitted disease
* Women who had received any hormone therapy for less than 60 days preceding the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 1 month
  Number of clinical pregnancy rate divided by the number of couples in which embryo transfer was performed

CONTACTS AND LOCATIONS:
Overall Officials: Edson Borges Jr., MD., PhD, Principal Investigator — Sapientiae Institute
Locations (1):
- Sapientiae Institute, São Paulo, São Paulo, Brazil